CLINICAL TRIAL: NCT07262229
Title: Self-management Digital Intervention to Promote Physical Activity in People Living With Chronic Obstructive Pulmonary Disease: a Pilot Randomized Controlled Trial Study Protocol
Brief Title: Self-management Digital Intervention to Promote Physical Activity in People Living With COPD
Acronym: Respir'airBPCO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut et Haute Ecole de la Santé la Source (Other)
Responsible Party: Principal Investigator, Ricardo Salgado, Senior Lecturer UAS, Institut et Haute Ecole de la Santé la Source
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Respir'air BPCO
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Self-management; E-health
Keywords: self-management; COPD; eHealth; digital intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Traditional pulmonologist follow-up, along with physiotherapy sessions
- Respir'air BPCO (Experimental): Self-management digital intervention (Respir'air BPCO)
  Interventions: Behavioral: Respir'air BPCO

INTERVENTIONS:
Behavioral: Respir'air BPCO — Self-management digital intervention (Respir'air BPCO) grounded in theory (Self-Care Theory of Chronic Illness, Self-Determination Theory of Human Motivation, and the Behavior Change Techniques taxonomy). The mobile application includes educational resources (text, video, images), examples of physical activities (walking, etc), environmental data (air quality), a personal activity log (daily steps), reminders and motivational messages.
  Arms: Respir'air BPCO

SUMMARY:
The goal of this pilot randomized controlled trial is to evaluate the feasibility, acceptability, and preliminary effects of a theory-based self-management digital intervention (Respir'air BPCO) designed to promote physical activity in patients with Chronic Obstructive Pulmonary Disease (COPD) after completion of a pulmonary rehabilitation program.

The main question it aims to answer is:

Is the Respir'air BPCO intervention (mobile app) feasible, acceptable, and preliminarily effective in increasing physical activity, enhancing self-management, improving motivation, and quality of life, while reducing dyspnea severity, exacerbations, and hospitalizations, compared with no additional intervention?

Researchers will compare an experimental group (receiving the Respir'air BPCO intervention + usual care) to a control group (no additional intervention, only usual care)

Participants will:

Be assigned either to the control group, receiving no additional intervention beyond usual care (traditional pulmonologist follow-up), or to the experimental group, receiving access to the Respir'air BPCO mobile app in addition to usual care.

* Complete baseline assessments immediately after finishing their in-person pulmonary rehabilitation program.
* Complete follow-up assessments at 3 months and 6 months after the start of the intervention

ELIGIBILITY:
Inclusion Criteria:

1. a GOLD COPD diagnosis stage 1 to 4, classification B or E;
2. admitted electively at Hospital for PR;
3. had completed the pulmonary rehabilitation program;
4. age over 18 years;
5. ability to provide informed consent;
6. internet access;
7. ownership of a smartphone or tablet;
8. self-assessed perceived ease of use of digital devices.

Exclusion Criteria:

1. clinical instability confirmed by the team of healthcare professionals;
2. severe cardiovascular disease confirmed by medical diagnosis;
3. recent history of neoplasia or autoimmune disease; other physical activity-limiting clinical condition confirmed by medical diagnosis (e.g. neurological disease);
4. other respiratory disease as primary diagnosis; e) inability to read, understand or speak French;

f) cognitive impairment diagnosed by the medical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Time required to complete recruitment | T0 - End of face-to-face PR program (Researchers expect to need 3 months to recruit 50 participants.)
Feasibility - The amount of missing data in the completed questionnaires | T0: Within 72 hours after completion of the face-to-face PR program T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
Feasibility - Potential refinements after the completion of the pilot study | From the start of the intervention to study completion, assessed for up to 9 months.
  A digital logbook for researchers' use, to record any observations or comments (patients and/or researchers perspectives) regarding the intervention design, content and/or usage, with the aim of informing potential refinements after the completion of the pilot study
Feasibility - Number of technical problems auto reported by the patient | T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
Feasibility - Intervention fidelity | T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  Exposure rate to all content available within the mobile application
Acceptability - Consent and retention rates | T -1: 1 week before completion of the face-to-face PR program (±72 hours)
  Consent rate: proportion of eligible participants who sign the informed consent form Retention rate: proportion of enrolled participants who remain in the study until the final assessment point
Acceptability - Acceptance rate of the allocated group | T -1: 1 week before completion of the face-to-face PR program (±72 hours)
  Acceptance rate will be assessed using administrative study records. It will be defined as the proportion of enrolled participants who agree to participate in the group to which they were allocated (control or intervention) immediately after randomization.
Acceptability - Rate of participants successfully recruited | T0: Within 72 hours after completion of the face-to-face PR program
Acceptability - Intervention acceptance | T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  Daily App Login Status
Acceptability - Intervention acceptance | T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  French-adapted version of the Treatment Acceptance and Preference (TAP) questionnaire.Responses are scored on a five-point Likert scale ranging from 0 ("not at all") to 4 ("extremely"), with higher scores reflecting greater acceptance.

SECONDARY OUTCOMES:
Preliminary effectiveness measures - Main variable: number of daily steps | T0: Within 72 hours after completion of the face-to-face PR program T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  Yamax Power Walker EX-510 pedometer over 5 consecutive days
Preliminary effectiveness measures - secondary variable: Self-management | T0: Within 72 hours after completion of the face-to-face PR program T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  Self-Care in Chronic Obstructive Pulmonary Disease Inventory (SC-COPDI). Overall standardized scores ranges for each of the three subscales range from 0 to 100. Higher scores indicate higher levels of self-care in COPD patients.
Preliminary effectiveness measures - secondary variable: Motivational regulation of physical activity | T0: Within 72 hours after completion of the face-to-face PR program T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  French-version of the Behavioural Regulation in Exercise Questionnaire-3 (BREQ-3). The score is obtained by averaging responses on a Likert scale ranging from "not at all true" (0) to "very true" (4). Higher scores indicate higher levels of motivation corresponding to the factor being assessed.
Preliminary effectiveness measures - secondary variable: Health-related quality of life | T0: Within 72 hours after completion of the face-to-face PR program T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  French version of the disease-specific St George's Respiratory Questionnaire. Each item is assigned a weight based on the level of distress attributed to each symptom or condition described. Overall scores range from 0 (no effect on quality of life) to a maximum score of 100 (maximum perceived suffering). A higher score means a poorer quality of life.
  French version of the EQ-5D-5L questionnaire. Each dimension is rated according to five levels of severity: from "no problem" (0) to "extreme problem" (4). EQ-5D-5L includes a visual analog scale (VAS) that allows participants to rate their general state of health on a scale from 0 to 100. Higher scores correspond to better health-related quality of life
Preliminary effectiveness measures - secondary variable: severity of dyspnea | T0: Within 72 hours after completion of the face-to-face PR program T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  French version of the mMRC Dyspnoea Scale. Uses a scale from 0 to 4. A score of 4 represents the highest severity of the dyspnea
Preliminary effectiveness measures - secondary variable: number of exacerbations | T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  Self-reported data
Preliminary effectiveness measures - secondary variable: number of hospitalizations | T1: 3 months after the start of the intervention (±1 week) T2: 6 months after the start of the intervention (±1 week)
  Self-reported data

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Salgado, MSc, Principal Investigator — Institut et Haute Ecole de la Santé la Source
Locations (1):
- Pôle de pneumologie de l'Hôpital de Rolle, Rolle, Switzerland